CLINICAL TRIAL: NCT01569243
Title: Using Activity Monitoring and Text Messaging For Behavior Change in a Diabetes Self-Management Program
Brief Title: Text to Move (TTM)Study
Acronym: TTM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: McKesson Foundation (Other)
Responsible Party: Principal Investigator, Joseph C. Kvedar, Dermatologist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2011-P-002708/1; MGH
Record Dates: First submitted 2012-03-28; First posted 2012-04-03 (Estimated); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes mellitus; Text messaging; Physical activity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care group (Other): Subjects in this group will receive the usual standard of care available at MGH.
  Interventions: Other: Usual care
- Text messaging group (Experimental): Subjects in this group will be enrolled to receive text messages aimed at providing bite-sized coaching based on measured step count to help improve activity levels and providing reminder, educational and motivation messages aimed at helping patients to meet their diabetes self-management goals.
  Interventions: Other: Text messages

INTERVENTIONS:
Other: Text messages — * Participants will receive diabetic medical care as usual.
  * Participants will be given an ActiHealth pedometer to measure daily activity.
  * In addition, they will be enrolled to receive the study text messages.
  Other Names: SMS
  Arms: Text messaging group
Other: Usual care — * Participants will receive diabetic medical care as usual.
  * In addition, participants in the control group will be given an ActiHealth pedometer to measure daily activity (step counts will be used as a proxy for activity).
  Other Names: Control
  Arms: Usual care group

SUMMARY:
This study is a 2-arm randomized controlled trial examining the effect of personalized text messages on physical activity and clinical outcomes in patients with type 2 diabetes mellitus.

The investigators hypothesize that:

i. The use of personalized text messages will promote physical activity in patients with T2DM.

ii. Increased physical activity and behavior change correlate with better clinical outcomes (Change in HbA1c).

iii. The text messaging program will lead to sustained physical activity behavior change in patients with T2DM

DETAILED DESCRIPTION:
Patients are referred into a Diabetes Self-Management Education (DSME) Support Program at Massachusetts General Hospital by a primary care provider at the time of diagnosis or as needed to gain better knowledge, awareness and understanding of their disease. Majority of the patients in the DSME program experience favorable outcomes; however, in key areas of T2DM management such as physical activity and nutrition, fewer patients experience success with their behavior goals, owing to the higher level of motivation required, and our inability to provide more frequent individually tailored feedback and coaching. In addition, we have observed that patients' behavior change is not sustained over time after finishing the DSME program.

In the proposed study, the investigators intend to augment DSME's evidence-based approach with two key connected health cornerstones - objective data collection and targeted personalized feedback. Using these two tools, we hypothesize that patients will be able to acquire new behaviors much sooner than status quo, and also maintain them for longer. Also, the scalability of the mobile component of the innovation will help us offer this evidence-based program to a much larger pool of patients, contributing greatly to the overall quality of diabetes management at our hospital.

The research team at Center for Connected Health will recruit participants from a pool of patients with T2DM who are participating in or who have gone through the DSME program at MGH Chelsea, MGH Revere or MGH Charlestown. These practices represent the most medically under served areas and serve low-income population. All of these practices have received recognition from the American Diabetes Association as having high-quality diabetes self-management education programs that meet the National Standards for Diabetes Self-Management Education.

120 participants will be enrolled and randomly assigned to one of the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Adults over the age of 18 years.
* HbA1c over 7.0%
* Patients with a diagnosis of T2DM at MGH Chelsea, MGH Revere MGH Charlestown or MGH Everett will be offered enrollment in the study.
* Must be willing to attend initial and close-out study visits
* Willingness to receive a maximum of 60 text messages/month for 6 months on their personal cellular phone.
* PC computer with internet access
* Fluency in English or Spanish (spoken and written)

Exclusion Criteria:

* Disability, medical or surgical condition preventing or precluding moderate physical activity.
* Significant cognitive deficits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2012-06; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
physical activity | 6 months
  Physical activity will be assessed by step counts measured by an ActiHealth pedometer and compared between the study arms.

SECONDARY OUTCOMES:
Clinical outcome | over 6 months (Day 1 and day 180)
  Will be assessed by pre and post HbA1c measurements
Change in physical activity behaviors | 6 months
  This will be assessed by Pre and post stage of behavior change based on the Stages of Motivational Readiness for Change model of the TTM.
Satisfaction with the program | 6 months
  This will be assessed using standardized Questionnaires at closeouts
Engagement to program | 6 months
  This will be measure quantitatively by:
  * number of days participant wore their pedometers in the study;
  * number of logins to the ActiHealth step count web portal;
  * percentage of messages a user responds to, in 2-way text messages

CONTACTS AND LOCATIONS:
Overall Officials: Kamal Jethwani, MD, MPH, Principal Investigator — Center for Connected Health
Locations (2):
- United States (2):
  - Center for Connected Health, Boston, Massachusetts
  - Partners Healthcare Center for Connected Health, Boston, Massachusetts

REFERENCES:
- [Background] Gibson TB, Song X, Alemayehu B, Wang SS, Waddell JL, Bouchard JR, Forma F. Cost sharing, adherence, and health outcomes in patients with diabetes. Am J Manag Care. 2010 Aug;16(8):589-600. PMID 20712392
- [Background] Funnell MM, Brown TL, Childs BP, Haas LB, Hosey GM, Jensen B, Maryniuk M, Peyrot M, Piette JD, Reader D, Siminerio LM, Weinger K, Weiss MA. National standards for diabetes self-management education. Diabetes Care. 2009 Jan;32 Suppl 1(Suppl 1):S87-94. doi: 10.2337/dc09-S087. No abstract available. PMID 19118294
- [Background] Watson AJ, Grant RW, Bello H, Hoch DB. Brave new worlds: how virtual environments can augment traditional care in the management of diabetes. J Diabetes Sci Technol. 2008 Jul;2(4):697-702. doi: 10.1177/193229680800200422. PMID 19885247
- [Background] Watson AJ, Bell AG, Kvedar JC, Grant RW. Reevaluating the digital divide: current lack of internet use is not a barrier to adoption of novel health information technology. Diabetes Care. 2008 Mar;31(3):433-5. doi: 10.2337/dc07-1667. Epub 2007 Dec 4. No abstract available. PMID 18056885
- [Background] Jethwani KS, Chandwani HS. The internet: revolutionizing medical research for novices and virtuosos alike. J Postgrad Med. 2008 Jan-Mar;54(1):49-51. doi: 10.4103/0022-3859.39194. No abstract available. PMID 18296809
- [Background] Watson AJ, Kvedar JC, Rahman B, Pelletier AC, Salber G, Grant RW. Diabetes connected health: a pilot study of a patient- and provider-shared glucose monitoring web application. J Diabetes Sci Technol. 2009 Mar 1;3(2):345-52. doi: 10.1177/193229680900300216. PMID 20144366
- [Background] Kulshreshtha A, Kvedar JC, Goyal A, Halpern EF, Watson AJ. Use of remote monitoring to improve outcomes in patients with heart failure: a pilot trial. Int J Telemed Appl. 2010;2010:870959. doi: 10.1155/2010/870959. Epub 2010 May 19. PMID 20508741
- [Background] Watson AJ, Bergman H, Williams CM, Kvedar JC. A randomized trial to evaluate the efficacy of online follow-up visits in the management of acne. Arch Dermatol. 2010 Apr;146(4):406-11. doi: 10.1001/archdermatol.2010.29. PMID 20404229
- [Derived] Horner GN, Agboola S, Jethwani K, Tan-McGrory A, Lopez L. Designing Patient-Centered Text Messaging Interventions for Increasing Physical Activity Among Participants With Type 2 Diabetes: Qualitative Results From the Text to Move Intervention. JMIR Mhealth Uhealth. 2017 Apr 24;5(4):e54. doi: 10.2196/mhealth.6666. PMID 28438728